CLINICAL TRIAL: NCT06217523
Title: Designing Therapy to Suit You - Personalised Hyperlipidaemia Therapies Guided by Pharmacogenomics (DTSY Lipid PGx): A Randomised Controlled Trial
Brief Title: Personalised Hyperlipidaemia Therapies Guided by Pharmacogenomics
Acronym: LipidPgx
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Singapore (Other)
Collaborators: Collabring Pte Ltd (Industry)
Responsible Party: Principal Investigator, Tan Su-Yin Doreen, Associate Professor, National University of Singapore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023/00280
Record Dates: First submitted 2023-11-06; First posted 2024-01-22 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Doctor-only care; receiving standard care without genetic information
- Intervention Group (Experimental): Pharmacist-guided care; dosing of statin medication based on genetic information
  Interventions: Other: Pharmacogenomics-directed Hyperlipidaemia Management

INTERVENTIONS:
Other: Pharmacogenomics-directed Hyperlipidaemia Management — Pharmacogenomics-directed Hyperlipidaemia Management
  Arms: Intervention Group

SUMMARY:
This trial aims to evaluate the impact of clinical pharmacists' pharmacogenomics-guided choice and statin titration for managing hyperlipidaemia.

The central hypotheses of this trial are (1) clinical pharmacists' pharmacogenomics-guided choice and titration of statins will lead to a more significant reduction in LDL-c; (2) lower incidence of myopathies with the use of statins for hyperlipidaemia management over 12 months compared to usual care by doctors alone. Active follow-up and titration should occur over the first six months. However, the participants will be followed up to 12 months to confirm the sustained LDL level attainment.

DETAILED DESCRIPTION:
The primary aims are:

* The changes in Low-Density Lipoprotein cholesterol (LDL-c), total cholesterol, triglycerides (TG), and high-density lipoprotein cholesterol (HDL-c) levels, and
* The incidence of myopathies over 12 months.

The secondary aims include:

* Characterisation of the pharmacogenomic relationship between serum levels of statins (and their metabolites) with the changes in LDL-c levels and incidence of myopathies over six months
* Economic outcomes include but are not limited to the cost-effectiveness of pharmacogenomic testing in attaining LDL-c targets
* Change in health-related quality of life over 12 months is measured using the EuroQoL 5-Dimension 5-Level questionnaire

ELIGIBILITY:
Inclusion Criteria:

* Participants between 21 and 75 years old
* Participants who are planning to start on statin* medication or whose LDL-c goals have not been met, per Appendix B.
* Participants who are able to communicate in English, Chinese or Malay.

Participants who are planning to start or will be started on the following doses are eligible: atorvastatin 10-80 mg/day, rosuvastatin 10-40 mg/day, or simvastatin 10-40 mg/day within the last two to four weeks before enrolment

Exclusion Criteria:

* Participants who are statin-intolerant or in whom statins are contraindicated
* Participants on a statin dosing schedule of every other day (EOD)
* Participants administered on potent Cytochrome P450 3A4 (CYP3A4) or Cytochrome P450 2C9 (CYP2C9) or OATP inhibitors or inducers.
* Participants on evolocumab and alirocumab prior to enrolment
* Participants with documented diagnosis of psychiatric conditions
* Participants requiring palliative care, end-of-life care, or those with a life expectancy of less than one year
* Pregnant and lactating women
* Participants with complaints of myalgia or muscle weakness at baseline, before the commencement of statin
* Participants who are unable to swallow a whole statin tablet

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Changes in LDL-C, HDL-C, Total cholesterol, and Triglycerides | 12 months
  Changes in LDL-C, HDL-C, Total cholesterol, and Triglycerides over 12 months
Change in creatine kinase | 6 months
  Changes in creatine kinase from baseline to six months only if myopathy complaints were present.
Incidence of myopathy complaints | 6 months
  Incidence of myopathy complaints at 1-month, 3-month, and 6-month

SECONDARY OUTCOMES:
(Clinician or Prescriber) Adherence to recommendations | 6 months
  The proportion of patients whose statin dose was prescribed in adherence to SLCO1B1 and/or ABCG2 phenotype recommendations, the proportion of patients with lipid-lowering drug changes following phenotype results, retrospective exploratory analyses of emerging gene predictors of lipid-control and myopathy
Cost effectiveness analysis | 12 months
  Cost effectiveness analysis will be measured as total direct medical cost per disability-adjusted life year
Direct medical costs | 12 months
  Total direct medical costs measured in USD will be computed from consultation costs, laboratory costs, and visits to other healthcare professionals.
Healthcare utilisation | 12 months
  Healthcare utilisation will be measured as the number of visits over 12 months
Changes in health-related quality of life | 12 months
  Changes in health-related quality of life will be measured using the utility score derived from EQ-5D-5L over 12 months. An improvement in scores imply a better quality of life.
Changes to beliefs about medications | 12 months
  Drug-Associated Risk Tool (DART)-Beliefs about Medicines Questionnaire (BMQ) scores will be computed. It is expected for responses to become more favourable over time

CONTACTS AND LOCATIONS:
Overall Officials: Ying Xian Chua, Principal Investigator — National University Polyclinics